CLINICAL TRIAL: NCT07006909
Title: Hair Isotope Analysis for Early Cancer Detection
Acronym: HI-CARE
Status: Not yet recruiting | Type: Observational
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Gunter G C Kuhnle, Professor of Nutrition and Food Science, University of Reading
Other Study IDs: HI-CARE 01
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: cancer; hair; stable isotope ratio
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cancer is a major health challenge, and early detection is crucial for improving patient outcomes. Research has shown that cancer can alter the way the body processes nutrients. This study aims to explore whether these metabolic changes can be detected through a simple, non-invasive method: analysing hair. Hair grows slowly over time, potentially capturing subtle metabolic changes that occur during cancer development. By studying the nitrogen stable isotope composition in hair samples donated by individuals diagnosed with cancer, we aim to identify potential early markers of the disease. Participants will be asked to donate a small strand of hair, which will be analysed using a laboratory technique called Isotope Ratio Mass Spectrometry (IRMS). The findings from this study could contribute to new, non-invasive screening tools for early cancer detection.

ELIGIBILITY:
Inclusion Criteria:

Cancer diagnosis, sufficient hair

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients in the UK
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2030-05-30 (Estimated); Study Completion 2030-05-30 (Estimated)

PRIMARY OUTCOMES:
longitudinal changes in d15N in hair | Approximately one year
  Longitudinal changes in d15N in hair samples to obtain a time-series

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participation will be anonymous